CLINICAL TRIAL: NCT01085617
Title: A Randomized Trial for Adults with Newly Diagnosed Acute Lymphoblastic Leukemia
Brief Title: Standard Chemotherapy with or Without Nelarabine or Rituximab in Treating Patients with Newly Diagnosed Acute Lymphoblastic Leukemia
Acronym: UKALL14
Status: Completed | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000667211; UCL-08-0167 (Other: UCL); EU-21009 (Other: NK); 2009-012717-22 (EudraCT Number); UCL-UKALL14 (Other: UCL); MREC-09-H0711-90 (Other: Research Ethics Committee); NCRI-UCL-08-0167 (Other: NK); CRUK-C27995-A9609 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Leukemia; Mucositis; Oral Complications
Keywords: oral complications; mucositis; untreated adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; Philadelphia chromosome positive adult precursor acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Mucositis | interventions — Fibroblast Growth Factor 7; Rituximab; Cyclophosphamide; Cytarabine; Daunorubicin; Etoposide; fludarabine phosphate; Imatinib Mesylate; Melphalan; Mercaptopurine; Methotrexate; nelarabine; pegaspargase; Vincristine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- B1 - Standard therapy (Active Comparator): Standard chemotherapy for precursor B-cell ALL
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: fludarabine phosphate; Drug: imatinib mesylate; Drug: melphalan; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate
- B2 - Rituximab (Experimental): Standard chemotherapy for precursor B-cell ALL plus weekly rituximab infusions during phase 1 induction
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: fludarabine phosphate; Drug: imatinib mesylate; Drug: melphalan; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate
- T1 - Standard therapy (Active Comparator): Standard chemotherapy for T-cell ALL
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: fludarabine phosphate; Drug: melphalan; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate
- T2 - Nelarabine (Experimental): Standard chemotherapy for T-cell ALL plus an additional course of treatment with nelarabine following phase 2 induction
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: fludarabine phosphate; Drug: melphalan; Drug: mercaptopurine; Drug: methotrexate; Drug: nelarabine; Drug: pegaspargase; Drug: vincristine sulfate
- P1 - standard palifermin (Active Comparator): 6 doses of palifermin before/after myeloablative stem cell transplant (randomisation closed due to lack of clinical relevance in 2016)
  Interventions: Biological: palifermin; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: total-body irradiation
- P2 - collapsed palifermin (Experimental): 1 x large dose of palifermin before myeloablative stem cell transplant and 3 low doses after transplant (randomisation closed due to lack of clinical relevance in 2016)
  Interventions: Biological: palifermin; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: palifermin
  Arms: P1 - standard palifermin; P2 - collapsed palifermin
Biological: rituximab
  Arms: B2 - Rituximab
Drug: cyclophosphamide
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: cytarabine
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: daunorubicin hydrochloride
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: etoposide
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: fludarabine phosphate
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: imatinib mesylate
  Arms: B1 - Standard therapy; B2 - Rituximab
Drug: melphalan
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: mercaptopurine
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: methotrexate
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: nelarabine
  Arms: T2 - Nelarabine
Drug: pegaspargase
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Drug: vincristine sulfate
  Arms: B1 - Standard therapy; B2 - Rituximab; T1 - Standard therapy; T2 - Nelarabine
Procedure: allogeneic hematopoietic stem cell transplantation
  Arms: P1 - standard palifermin; P2 - collapsed palifermin
Radiation: total-body irradiation
  Arms: P1 - standard palifermin; P2 - collapsed palifermin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known which regimen of combination chemotherapy given together with or without monoclonal antibodies is more effective in treating patients with newly diagnosed acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is studying standard chemotherapy to see how well it works when given together with or without rituximab, and with or without nelarabine in treating patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the addition of a monoclonal antibody (none vs. rituximab) improves event-free survival (EFS) in patients with newly diagnosed precursor B-cell acute lymphoblastic leukemia (ALL).
* To determine if the addition of nelarabine improves outcome for patients with T-cell ALL.

Secondary

* To determine the tolerability of pegaspargase in induction therapy of all patients.
* To compare anti-asparaginase antibody levels in patients with B-lineage ALL.
* To determine whether risk-adapted introduction of unrelated donor hematopoietic stem cell transplantation (HSCT) (myeloablative conditioning in patients ≤ 40 years old and non-myeloablative conditioning in patients > 40 years old) results in greater EFS for patients at highest risk of relapse.
* To compare the efficacy of two schedules (standard vs collapsed) of palifermin in preventing severe mucosal toxicity in patients treated with etoposide, total-body irradiation, and HSCT-conditioning therapy.
* To assess the late effects of this treatment in these patients.
* To identify and describe some of the adverse physical and psychosocial consequences of this disease and its treatment.

OUTLINE: This is a multicenter study. There are 3 randomizations at different timepoints in the trial, each patient undergoes at least 1 but no more than 2 randomizations.

* Part 1 standard induction therapy (all patients*, weeks 1-4): Patients receive daunorubicin hydrochloride IV over 20 minutes and vincristine sulfate IV over 5-10 minutes on days 1, 8, 15, and 22; oral dexamethasone once a day on days 1-5, 8-11, and 15-18; pegaspargase IV over 1-2 hours on days 4 and 18; and methotrexate intrathecally (IT) on day 14.

NOTE: *Patients with Philadelphia-positive (Ph+) disease should also receive oral imatinib mesylate once a day on days 1-28.

* Randomized concurrent monoclonal antibody therapy (for patients with precursor B-cell acute lymphoblastic leukemia [ALL]): Patients with precursor B-cell ALL are randomized to 1 of 4 monoclonal antibody treatment arms (given concurrently with part 1 standard induction therapy):

  * Arm B1: Patients do not receive any monoclonal antibody therapy.
  * Arm B2 : Patients receive rituximab IV on days 3, 10, 17, and 24.

    * Part 2 standard induction therapy (all patients*, weeks 5-8): Patients receive cyclophosphamide IV over 30 minutes on days 1 and 15; cytarabine IV on days 2-5, 9-12, 16-19, and 23-26; oral mercaptopurine once a day on days 1-28; and methotrexate IT on days 1, 8, 15, and 22.

NOTE: *Patients with Ph+ disease should also receive oral imatinib mesylate once a day on days 1-30.

* Randomized subsequent nelarabine therapy (for Patients with T-cell ALL) Patients with T-cell ALL are randomized to 1 of 2 treatment arms, to be administered after completion of part 2 standard induction therapy.

  * Arm T1: Patients do not receive any other therapy during induction.
  * Arm T2: Patients receive nelarabine IV over 2 hours on days 1, 3, and 5. Patients who do not achieve complete remission (CR) after part 2 standard induction therapy are taken off study.

    * Intensification/central nervous system prophylaxis (patients not eligible for transplant OR patients > 40 years at study entry and eligible for transplant)*: Beginning after recovery from part 2 standard induction therapy, patients receive high-dose methotrexate IV on days 1 and 15 and pegaspargase IV over 1-2 hours on days 2 and 16.

NOTE: *Patients with Philadelphia-positive (Ph+) disease should also receive oral imatinib mesylate once a day on days 1-28.

Patients eligible for allogeneic hematopoietic stem cell transplantation (HSCT) (i.e., any patient with an HLA-compatible sibling donor or high risk patients with a molecularly matched donor) undergo transplantation; patients not eligible for HSCT undergo consolidation followed by maintenance therapy.

* Consolidation therapy* (patients not eligible for transplantation):

  * Course 1: Beginning after completion of intensification therapy, patients receive cytarabine IV and high-dose etoposide IV over 30 minutes on days 1-5, pegaspargase IV over 1-2 hours on day 5, and methotrexate IT on day 1. Patients proceed to course 2 beginning 3 weeks after the start of course 1 or when neutrophils recover.
  * Course 2: Patients receive cytarabine IV and high-dose etoposide IV over 30 minutes on days 1-5 and methotrexate IT on day 1. Patients proceed to course 3 beginning 3 weeks after the start of course 2 or when neutrophils recover.
  * Course 3 (delayed intensification): Patients receive daunorubicin hydrochloride IV over 20 minutes and vincristine sulfate IV over 5-10 minutes on days 1, 8, 15, and 22; pegaspargase IV over 1-2 hours on day 4; oral dexamethasone once a day on days 1-4, 8-11, 15-18, and 22-25; methotrexate IT on days 2 and 17; cyclophosphamide IV on day 29; cytarabine IV on days 30-33 and 37-40; and oral mercaptopurine once a day on days 29-42. Patients proceed to course 4 after neutrophils recover.
  * Course 4: Patients receive cytarabine IV, high-dose etoposide IV, and methotrexate IT as in course 2.

NOTE: *Patients with Ph+ disease should also receive oral imatinib mesylate once a day on days 1-7 in courses 1 and 2, on days 2-42 in course 3, and on days 1-8 in course 4.

* Maintenance therapy (patients not eligible for transplantation): Patients receive vincristine sulfate IV every 3 months, oral prednisolone once a day on days 1-5 every 3 months, oral mercaptopurine once daily, methotrexate IV or orally once a week, and methotrexate IT every 3 months for 2 years.
* Transplant conditioning and allogeneic HSCT:

  * Myeloablative-conditioning and allogeneic HSCT (patients ≤ 40 years old at study entry): Patients undergo total-body irradiation on days -7 to -4 and receive high-dose etoposide IV over 4 hours on day -3 or high-dose cyclophosphamide IV over 2 hours on days -3 and -2. Patients then undergo allogeneic HSCT on day 0.

Patients are stratified according to gender, donor (sibling donor vs. matched unrelated donor), and cellular type of ALL (precursor B-lineage vs. T-lineage). Patients are randomized to receive 1 of 2 palifermin treatment arms.

* Arm P1 (standard dose): Patients receive palifermin IV on days -3 to 2.
* Arm P2 (collapsed dose): Patients receive palifermin IV on days -1 to 2.

  * Non-myeloablative-conditioning and allogeneic HSCT (patients > 40 years old at study entry): Patients receive fludarabine phosphate IV over 30-60 minutes on days -7 to -3 and melphalan IV over 90 days on day -1. Recipients of unrelated donor HSCT also receive alemtuzumab IV over 2 hours on day -2 and -1; recipients of sibling HSCT receive alemtuzumab IV over 2 hours on day -1. Patients then undergo allogeneic HSCT on day 0. Patients also receive post transplant methotrexate IT every 3 months for 2 years.

Patients undergo blood and bone marrow sample collection periodically for correlative studies.

After completion of study treatment, patients are followed annually.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed, previously untreated acute lymphoblastic leukemia

  * A pre-phase steroid treatment of 5-7 days is required and can be started prior to registration
* Philadelphia chromosome-negative or -positive patients are eligible
* No blast transformation of chronic myeloid leukemia
* No mature B-cell leukemia [i.e., Burkitt disease t(8,14)(q24 ;q32)] or variant c-myc translocations [e.g., t(2;8)(p12;q24), t(8;22)(q24;q11)]
* Patients who undergo study transplantation must have HLA-compatible sibling or unrelated donor

  * 8/8 molecular match at -A, -B, -C, and -DR (DQ mismatch is permitted)
* Patients meeting ≥ 1 the following criteria are considered high-risk:

  * Over 40 years old
  * WBC ≥ 30 x 10^9/L (precursor-B) OR ≥ 100 x 10^9/L (T-lineage)
  * Any 1 or more of the following cytogenetic abnormalities:

    * t(4;11)(q21;q23)/MLL-AF4
    * Low hypodiploidy/near triploidy (30-39 chromosomes/60-78 chromosomes)
    * Complex karyotype (≥ 5 chromosomal abnormalities)
    * Philadelphia chromosome t(9;22) (q34;q11)/BCR-ABL1 (detected by cytogenetic or molecular methods)
  * High-risk minimal-residual disease after completion of part 2 standard induction therapy

PATIENT CHARACTERISTICS:

* No known HIV infection
* Not pregnant or nursing (no nursing during and for 12 months after completion of study therapy)
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 12 months after completion of study therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-12 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 3 years
  Time from randomisation to relapse or death from any cause

SECONDARY OUTCOMES:
Anti-asparaginase antibodies in patients treated with monoclonal antibody therapy | Throughout treatment
  Antibody levels in sequential samples during pegylated asparaginase treatment
Overall survival | 3 years
  Time from randomisation to death from any cause
Complete remission (CR) rate | Throughout treatment
  Proportion of patients achieving morphological complete remission
Minimal-residual disease quantification after first phase of induction and post-transplantation | Throughout treatment
  Minimal residual disease measured at central laboratory after phase 1 induction and post transplant
Relapse rate (including bone marrow and CNS relapse) | 3 years
  Proportion of patients experiencing a bone marrow of CNS relapse after entering complete remission
Death in CR | 3 years
  Proportion of patients dying while their ALL is in complete remission
Toxicity related to pegaspargase | Throughout treatment
  Rates of hypersensitivity, changes to Erwinia, or withdrawal of asparaginase treatment
Mucositis score in patients treated with palifermin | 30 days
  OMQD score, number of doses of methotrexate given, acute GVHD rates

CONTACTS AND LOCATIONS:
Overall Officials: Adele K. Fielding, Principal Investigator — University of York

REFERENCES:
- [Derived] Marks DI, Clifton-Hadley L, Copland M, Hussain J, Menne TF, McMillan A, Moorman AV, Morley N, Okasha D, Patel B, Patrick P, Potter MN, Rowntree CJ, Kirkwood AA, Fielding AK. In-vivo T-cell depleted reduced-intensity conditioned allogeneic haematopoietic stem-cell transplantation for patients with acute lymphoblastic leukaemia in first remission: results from the prospective, single-arm evaluation of the UKALL14 trial. Lancet Haematol. 2022 Apr;9(4):e276-e288. doi: 10.1016/S2352-3026(22)00036-9. PMID 35358442
- [Derived] Marks DI, Kirkwood AA, Rowntree CJ, Aguiar M, Bailey KE, Beaton B, Cahalin P, Castleton AZ, Clifton-Hadley L, Copland M, Goldstone AH, Kelly R, Lawrie E, Lee S, McMillan AK, McMullin MF, Menne TF, Mitchell RJ, Moorman AV, Patel B, Patrick P, Smith P, Taussig D, Yallop D, Alapi KZ, Fielding AK. Addition of four doses of rituximab to standard induction chemotherapy in adult patients with precursor B-cell acute lymphoblastic leukaemia (UKALL14): a phase 3, multicentre, randomised controlled trial. Lancet Haematol. 2022 Apr;9(4):e262-e275. doi: 10.1016/S2352-3026(22)00038-2. PMID 35358441
- [Derived] Mitchell RJ, Kirkwood AA, Barretta E, Clifton-Hadley L, Lawrie E, Lee S, Leongamornlert D, Marks DI, McMillan AK, Menne TF, Papaemmanuil E, Patel B, Patrick P, Rowntree CJ, Zareian N, Alapi KZ, Moorman AV, Fielding AK. IKZF1 alterations are not associated with outcome in 498 adults with B-precursor ALL enrolled in the UKALL14 trial. Blood Adv. 2021 Sep 14;5(17):3322-3332. doi: 10.1182/bloodadvances.2021004430. PMID 34477813
- [Derived] Patel B, Kirkwood AA, Dey A, Marks DI, McMillan AK, Menne TF, Micklewright L, Patrick P, Purnell S, Rowntree CJ, Smith P, Fielding AK. Pegylated-asparaginase during induction therapy for adult acute lymphoblastic leukaemia: toxicity data from the UKALL14 trial. Leukemia. 2017 Jan;31(1):58-64. doi: 10.1038/leu.2016.219. Epub 2016 Aug 2. PMID 27480385